CLINICAL TRIAL: NCT04989998
Title: A Prospective, Multi-center, Randomized Controlled Study to Evaluate Patient Outcomes Using Hip7 Software as Compared to Conventional Surgical Technique in S+N Total Hip Arthroplasties (THA)
Brief Title: Patient Outcomes Using HIP7 Software as Compared to Conventional THA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: update to marketing strategy for hip robotics and related instrumentation
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIP7.2020.10
Record Dates: First submitted 2021-06-28; First posted 2021-08-04 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Hip Replacement
Keywords: HIP7; Total Hip Arthroplasties (THA)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Hip7 Software on Kick/ CORI platforms (Experimental): Subjects will receive total hip arthroplasty surgery using Hip7 on Kick or CORI platform utilizing R3 Polarstem implants.
  Interventions: Device: Hip7 Software on Kick/ CORI platforms
- Conventional procedures with standard, manual instrumentation and digital templating techniques (Active Comparator): Subjects will receive total hip arthroplasty surgery using conventional procedures with standard instrumentation and digital templating techniques utilizing R3 Polarstem implants.
  Interventions: Device: Conventional surgical procedures

INTERVENTIONS:
Device: Hip7 Software on Kick/ CORI platforms — Total hip arthroplasty surgery using Hip7 software on Kick or CORI platforms using R3 Polarstem implants.
  Arms: Hip7 Software on Kick/ CORI platforms
Device: Conventional surgical procedures — THA surgery using standard, manual instrumentation and digital templating techniques using R3 polarstem implants.
  Arms: Conventional procedures with standard, manual instrumentation and digital templating techniques

SUMMARY:
The study is designed to demonstrate how Hip7 software can lead to improved patient outcomes compared to conventional procedures with standard instrumentation for total hip arthroplasties (THA) surgery.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, randomized, controlled clinical study in total hip arthroplasties (THA) surgery. The subjects meeting the inclusion/exclusion criteria specified in the protocol will receive THA using either Hip7 software or conventional instrumentation.

The clinical follow-up evaluation will be performed preoperatively (Baseline), operatively, 6 weeks, 6 and 12 months after surgery using patient reported outcome measures regarding their general health, hip and physical abilities, quality of life and pain level.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or legal guardian must provide written informed consent (reference section 7.5).
2. Subjects eighteen (18) years or older and considered skeletally mature.
3. Willing and able to make all required study visits.
4. Able to follow instructions and deemed capable of completing the FJS, OHS, HOOS and EQ-5D-5L questionnaires.
5. Subject requires a THA as a primary indication.
6. Subject is a suitable candidate for implanting specific S+N implant system in the investigator's judgement.
7. Subject agrees to consent to and to follow the study visit schedule (as defined in the study protocol and informed consent form), by signing the Ethics Committee (EC) approved informed consent form.
8. Subject plans to be available through 12 months postoperative follow-up
9. Routine radiographic assessment including CT and X-ray is possible.

Exclusion Criteria:

1. Contraindicated for robotic THA or POLAR3 hip implant.
2. Participation in the treatment period of another clinical trial within thirty (30) days of Visit 1, or during the study.
3. Women who are pregnant, nursing, or of child-bearing potential who are not utilizing highly effective birth control measures.
4. Any subject that meets the definition of a Vulnerable Subject per International Organization for Standardization (ISO) 14155:2011 Section 3.44.
5. Subjects who have participated previously in this trial through THA on their other hip.
6. Subjects with a history of poor compliance with medical treatment (i.e have mental illness, drug or alcohol addiction).
7. Subjects who need a THA procedure on the index joint as a revision for a previously failed surgery.
8. Subjects suspected to need bilateral surgery in the next 12 months.
9. Subject has received THA on the opposing hip within the previous 6 months.
10. Subjects not understanding the language used in the Informed Consent Form.
11. Subjects with an active infection or sepsis (treated or untreated).
12. Subjects morbidly obese with a BMI greater than 40.
13. Subjects in the opinion of the Investigator, has advanced osteoarthritis or joint disease at the time of surgery and are better suited for an alternate procedure.
14. Subjects that have condition(s) that may interfere with the THA survival or outcome (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease, or an active, local infection).
15. Subjects, in the opinion of the Investigator, has a neuromuscular disorder that prohibited control of the index joint.
16. Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Forgotten Joint Score (FJS) | 12 months post-surgery
  Compare Forgotten Joint Score (FJS) utilizing Hip7 software on Kick & CORI platforms with POLAR3 system to conventional procedures with standard instrumentation and digital templating techniques at 12 months post-operation. The FJS-12 Questionnaire comprises measures for assessment of joint-specific patient reported outcomes that focuses on subject's awareness of replaced joint in everyday life. Joint awareness defined as any unintended perception of a joint. Subjects rate awareness of their hip arthroplasty in 12 questions with a 5-point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". Scores are summed & linearly transformed in a 0-100 scale with a high value reflecting subject's ability to forget the replaced hip joint during daily living activities.

SECONDARY OUTCOMES:
Change in Frequency of Reduction of Outliers | 6 weeks post surgery
  Frequency of reduction of outliers* with Hip7 software as compared to conventional procedures (as defined by literature) using digital templating techniques for posterior and direct anterior approaches
  *Outliers are defined as acetabular component placement outside the desired "safe zone". Two most commonly used safe zones are described by Lewinnek and Callanan with the inclination and anteversion values outlined below: Callanan Safe Zone -- Anteversion between 5-25 degrees, Inclination between 30-45 degrees. Lewinnek - Anteversion between 5-25 degrees, Inclination between 30-50 degrees [i.e. 40° ± 10° and 15° ± 10°].
Patient Reported Outcomes: Hip Disability and Osteoarthritis Outcome Score (HOOS) | 12 months post-surgery
  The HOOS is developed as an instrument to assess the subject's opinion about their hip and associated problems. HOOS consists of 5 subscales: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and hip related QOL. The last week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Patient Reported Outcomes: Oxford Hip Score (OHS) | 12 months post-surgery
  The OHS is a 12-item questionnaire for patients who undergo total hip replacement (THR) to complete. Patients are asked to reflect on their pain and functional ability over the previous four weeks. There are two domains (pain and function) with six items or questions in each. Each item has four possible responses. Responses were from 1 = least difficult to 4= most difficult. Item scores are summed to give a total score from anywhere between 0 and 48. The lower the score, the better the outcome.
Patient Reported Outcomes: EuroQol (European Quality of Life) five-dimensional Five-level (EQ-5D-5L) | 12 months post-surgery
  The EQ-5D-5L questionnaire consists of two parts. Part one is the descriptive system to describe the subject's health state and consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The subject indicates their health state by marking the most appropriate statement in each of the 5 areas. Responses are converted to scores ranging from less than 0 to 1.0 with high scores representing higher health utility. Part two is the EQ Visual Analog Scale (VAS) that records the subject's self-rated health on a vertical visual analogue scale. Scale ranges from 0-100 with 100 labelled "The best health you can imagine" and 0 "The worst health you can imagine".
Cup placement accuracy | 6 weeks post-op
  To demonstrate cup placement accuracy (defined as the difference between inclination, anteversion, leg length, and offset target) from the Computerized Tomography [CT]).
Assess Pelvic Tilt at 6 Weeks | 6 weeks post-op
  A CT scan will assess pelvic tilt (angle of pelvic bone in relation to spine and femur)
Assess Range of Motion of Femur at 6 Weeks | 6 weeks post-op
  Medical staff will measure angles of femur movement in order to assess active range of motion. Active range of motion measures include angles of active flexion, abduction, adduction, external rotation and internal rotation.
Assess Frequency of Femur Head Dislocation at 6 Weeks | 6 weeks post-op
  Whether the subject experienced femoral head dislocation will be assessed at 6 weeks post op. Femoral head dislocation will be determined based on the count of participants with joint dislocation responses recorded by the investigator in the Adverse Events Case Report Form (CRF).

CONTACTS AND LOCATIONS:
Overall Officials: Edward T Davis, MB ChB, M.Sc, PGCME, FRCS(T&O), Principal Investigator — The Royal Orthopaedic Hospital NHS Foundation Trust; Yixin Zhou, Principal Investigator — Beijing Jishuitan Hospital

IPD SHARING:
Plan to Share IPD: No